CLINICAL TRIAL: NCT02512562
Title: A Phase-1, Open-label, Two Group, Fixed-Sequence Study to Evaluate the Effect of ACH-3102 and Simeprevir on AL-335 Pharmacokinetics in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of ACH-3102 and Simeprevir on AL-335 Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL-335-602
Record Dates: First submitted 2015-07-06; First posted 2015-07-31 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — adafosbuvir; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Group 1: AL-335, Simeprevir and ACH-3102 (Active Comparator): AL-335, ACH-3102, and Simeprevir dosed in healthy human volunteers once daily for 24 days.
  Interventions: Drug: AL-335; Drug: ACH-3102; Drug: Simeprevir
- Group 2: AL-335, Simeprevir and ACH-3102 (Active Comparator): AL-335, ACH-3102, and Simeprevir dosed in healthy human volunteers once daily for 24 days.
  Interventions: Drug: AL-335; Drug: ACH-3102; Drug: Simeprevir

INTERVENTIONS:
Drug: AL-335 — AL-335 is a prodrug being developed as an orally administered anti-HCV therapeutic.
Drug: ACH-3102 — ACH-3102 is an NS5A inhibitor being developed as an orally administered anti-HCV therapeutic.
Drug: Simeprevir — Simeprevir is an orally active, small molecule inhibitor of the NS3/4A protease of HCV and indicated for the treatment of chronic HCV infection as a component of a combination antiviral treatment regimen.
  Other Names: Olysio

SUMMARY:
This is an open-label, two-group, fixed-sequence study to evaluate the effect of ACH-3102 and Simeprevir on AL-335 pharmacokinetics in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written consent.
2. In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions and is likely to complete the study as planned.
3. Subject is in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests and ECG.
4. Male or female, 18-60 years of age.
5. Body mass index (BMI) 18-32 kg/m2, inclusive. The minimum weight is 50 kg. No more than 25% of subjects may be enrolled with a BMI ≥ 30 kg/m2.
6. A female subject is eligible to participate in this study if she is of non-childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females)). A post-menopausal female receiving hormone replacement therapy who is willing to discontinue hormone therapy 28 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation.
7. If male, subject is surgically sterile or practicing specific forms of birth control until 6 months after the end of the study. Males must agree to refrain from sperm donation from check-in through 6 months after dosing.
8. Willing to avoid prolonged sun exposure while taking SMV and through follow-up. Subjects should also be advised to use a broad spectrum sun screen and lip balm of at least sun protection factor (SPF) > 30 to help protect against potential sunburn.

Exclusion Criteria:

1. Pregnant or nursing (lactating) females, confirmed by a positive HCG laboratory test or females contemplating pregnancy. Men whose female partners are pregnant or contemplating pregnancy from the date of screening until 6 months after their last dose of study drugs.
2. Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid or any other medical illness or psychiatric disorder, as determined by the Investigator and/or Sponsor's Medical Monitor.
3. Positive screening test for hepatitis B, C or HIV serology. Subjects previously infected with HCV and achieved a sustained virologic response with treatment (no detectable HCV RNA 6 months post treatment) are eligible.
4. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements.
5. Participation in an investigational drug trial or having received an investigational vaccine within 30 days or 5 half-lives (whichever is longer) prior to study medication.
6. Clinically significant abnormal ECG findings. Particularly, a history or family history of prolonged QT syndrome (e.g., torsade de pointes) or sudden cardiac death.
7. ECG with PR > 200 ms, QRS > 120 ms, QTcF > 450 ms, as assessed by centrally read 12 lead ECG at the screening visit.
8. Clinically significant blood loss or elective blood donation of significant volume (i.e., > 500 mL) within 60 days of first dose of study drug; > 1 unit of plasma within 7 days of first dose of study drug.
9. Abnormal heart rate, respiratory rate, temperature or blood pressure values outside of the normal range (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest). One repeat measurement after an additional 5 minutes of rest is permitted.
10. Evidence of active infection.
11. Unwilling to abstain from alcohol for at least 1 week prior to the start of dosing through the study completion visit.
12. History of regular alcohol intake > 7 units per week of alcohol for females and > 14 units per week for males (one unit is defined as 10 g alcohol) within 3 months of the screening visit.
13. History of tobacco use or used nicotine-containing products within 3 months of the screening visit.
14. The subject has a positive pre-study drug screen.
15. The use of concomitant medications, including prescription, over the counter medications, herbal medications, inducers or inhibitors of CYP450 enzymes or drug transporters (including P-gp) within 14 days prior to the first dose of study medication is excluded, unless approved by the Sponsor's Medical Monitor. Occasional use of acetaminophen is permitted.
16. Exposure to more than four new investigational entities within 12 months prior to the first dosing day.
17. Hypersensitivity to the active substances or to any of the excipients of AL-335, ACH-3102 or SMV.
18. Subjects of East Asian ancestry.
19. Abnormal biochemistry or hematology laboratory results obtained at screening. Elevated bilirubin in subjects with suspected Gilbert's disease is allowed.
20. Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Multiple dose PK Profile, Cmax and AUC: effect of ACH-3102 on AL-335 and metabolites | From screening to Day 28 follow-up visit
  To evaluate the effect of multiple oral doses of ACH-3102, on the multiple oral dose PK of AL-335 and metabolites
Multiple dose PK Profile, Cmax and AUC: effect of Simeprevir on AL-335 and metabolites | From screening to Day 24 visit
  To evaluate the effect of multiple oral doses of Simeprevir, on the multiple oral dose PK of AL-335 and metabolites
Multiple dose PK Profile, Cmax and AUC: effect of ACH-3102 and Simeprevir on AL-335 and metabolites | From screening to Day 28 follow-up visit
  To evaluate the effect of multiple oral doses of ACH-3102 and Simeprevir, on the multiple oral dose PK of AL-335 and metabolites

SECONDARY OUTCOMES:
Safety Data: Composite number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG and abnormal clinical laboratory results | From screening to Day 28 follow-up visit
  Tabulation of the number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG and abnormal clinical laboratory results (including chemistry, hematology, and urine).
Steady-state PK Profile from Clast, t1/2, Tmax, Tlast, CL/F, Vz/F, λz: effect of AL-335 and ACH-3102 on Simeprevir | From screening to Day 28 follow-up visit
  To determine the potential effect of AL-335 and/or ACH-3102 on the steady-state PK of Simeprevir.
Steady-state PK Profile from Clast, t1/2, Tmax, Tlast, CL/F, Vz/F, λz: effect of AL-335 and Simeprevir on ACH-3102 | From screening to Day 28 follow-up visit
  To determine the potential effect of AL-335 and/or Simeprevir on the steady-state PK of ACH-3102.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Rennes, France

REFERENCES:
- [Derived] Valade E, Valenzuela B, Kakuda TN, Westland C, McClure MW, Ouwerkerk-Mahadevan S, Perez-Ruixo JJ, Ackaert O. Characterizing the Pharmacokinetic Interaction Between Simeprevir and Odalasvir in Healthy Volunteers Using a Population Modeling Approach. AAPS J. 2018 Oct 22;20(6):111. doi: 10.1208/s12248-018-0271-0. PMID 30350297
- [Derived] Kakuda TN, McClure MW, Westland C, Vuong J, Homery MC, Poizat G, Viguerie L, Denot C, Patat A, Zhang Q, Hui J, Apelian D, Smith DB, Chanda SM, Fry J. Pharmacokinetics, safety, and tolerability of the 2- and 3-direct-acting antiviral combination of AL-335, odalasvir, and simeprevir in healthy subjects. Pharmacol Res Perspect. 2018 Apr 30;6(3):e00395. doi: 10.1002/prp2.395. eCollection 2018 Jun. PMID 29736243